CLINICAL TRIAL: NCT06977308
Title: A Multimodal Imaging Study of Dopamine in Early Psychosis
Acronym: MISDEP
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Columbia University Irving Medical Centre (Unknown); Research Foundation for Mental Hygiene, Inc. / Columbia University (Unknown); Stony Brook Medicine (Unknown)
Responsible Party: Principal Investigator, Ragy Girgis, Professor of Clinical Psychiatry, New York State Psychiatric Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 8361; 1R01MH128330 (NIH)
Record Dates: First submitted 2025-05-08; First posted 2025-05-18 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Clinical High Risk for Psychosis (CHR)
Keywords: clinical high risk for psychosis
MeSH Terms: interventions — Methylphenidate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Methylphenidate (Experimental): Each subject will receive one oral dose of 60mg methylphenidate in between 2 PET scans with [11C]raclopride.
  Interventions: Drug: Methylphenidate (MPH); Drug: [11C]raclopride

INTERVENTIONS:
Drug: Methylphenidate (MPH) — Each participate will receive one oral dose of 60mg methylphenidate.
Drug: [11C]raclopride — This is the radiotracer that will be used along with methylphenidate to quantify dopamine transmission in this study. It is experimental and used for imaging purposes.

SUMMARY:
The development of new treatments for psychosis, a psychiatric condition that is prevalent and highly disabling despite antipsychotic medications, has been limited, in part, by a lack of information from brain imaging studies during the period that leads to the development of psychotic symptoms. In this project the investigators will use Positron Emission Tomography (PET) and neuromelanin-sensitive magnetic resonance imaging (NM-MRI) to examine a brain chemical that is involved in schizophrenia called dopamine and where it first becomes abnormal. The investigators will use multimodal PET/MR imaging (i.e., [11C]raclopride w/MPH challenge and NM-MRI) in the same CHR patients. The investigators will recruit 115 clinical high risk individuals. All subjects will undergo [11C]raclopride w/methylphenidate challenge and neuromelanin-MRI imaging along with clinical assessments. Patients will be followed every 3 months for two years or until conversion to psychosis, whichever comes first, to assess for conversion to psychosis and clinical outcomes.

DETAILED DESCRIPTION:
A large body of evidence suggests that abnormal striatal dopamine (DA) transmission is a key pathophysiological phenomenon in psychosis, mainly within the associative striatum (AST). However, it remains unclear where striatal DA abnormalities in psychosis start and whether they can be turned into a biomarker for development of psychotic illness. Early studies in individuals at clinical high-risk for psychosis (CHR) demonstrated that patients had higher [18F]DOPA uptake (i.e., DA synthesis capacity) in the AST compared to healthy control subjects (HC). One study reported that CHR individuals who developed a syndromal psychotic disorder had higher [18F]DOPA uptake than CHR individuals who did not progress. However, more recent work in larger samples has not replicated either finding. The investigators recently completed a feasibility study in which the investigators used [11C]-(+)-PHNO w/methylphenidate (MPH) challenge to examine intrasynaptic DA transmission in 14 CHR individuals and 14 HCs. The investigators found that intrasynaptic DA transmission was significantly elevated in the limbic/ventral striatum (VST), and not in any other ROI, in CHR individuals compared to HC. There was a strong correlation between intrasynaptic DA transmission in VST and total negative symptoms in the CHR group in which greater displacement was related to less negative symptoms. CHR subjects experienced no change in positive symptoms with MPH challenge, which demonstrates the safety of this technique. Additionally, our preliminary data with neuromelanin sensitive MRI (NM-MRI), a MR technique of measuring NM, a metabolite of DA, in different presynaptic nuclei (the substantia nigra [SN; the ventromedial portion of which projects to the AST] and ventral tegmental area [VTA; which projects to the VST]), demonstrate positive relationships between the contrast-to-noise ratio (CNR) of NM-MRI in the SN and positive symptoms in CHR and SCZ subjects. Taken together, these findings may reflect: 1) that striatal DA abnormalities in early psychosis progress in a temporo-spatial manner from VST to AST; 2) a clinical pattern in which negative symptoms are related to limbic DA transmission and positive symptoms reflect DA function in associative regions; 3) differences in biomarker (i.e., PHNO w/MPH challenge, NM-MRI, [18F]DOPA). This proposal will aim to advance the understanding of the nature, topography, and timing of striatal DA alterations in early psychosis by using multimodal PET/MR imaging (i.e., [11C]raclopride w/MPH challenge and NM-MRI) in the same CHR patients. The investigators will recruit 115 CHR individuals. All subjects will undergo [11C]raclopride w/MPH and NM-MRI imaging along with clinical assessments. Patients will be followed every 3 months for two years or until conversion to psychosis, whichever comes first, to assess for conversion to psychosis and clinical outcomes. Clarifying the nature, timing, and topography of DA abnormalities in early psychosis will greatly inform translational studies and could provide support for alternative initial therapeutic interventions to prevent progression in early psychosis.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females between 18 and 30 years old
2. Capacity to give informed consent
3. Clinical High Risk (i.e., APSS, GRDS, BIPS)
4. Antipsychotic free for 3 weeks before the PET scan
5. Clinically stable enough for the study

Exclusion Criteria:

1. Any substance use disorder, of any severity, within the previous month (before PET scan; not including nicotine or caffeine)
2. Any current use of substance of abuse besides THC/marijuana/cannabis/nicotine/caffeine (on day of PET only)
3. Daily tobacco use
4. Pregnancy
5. Lactation
6. Presence of insulin-dependent diabetes
7. IQ < 70 (i.e., WTAR < 6)
8. Acute risk for suicide (i.e., score of 4-5 within the previous month or 6 within the previous 3 months on the CSSRS) or violence, or history of severe violent behavior that may be exacerbated by methylphenidate
9. Presence of metallic objects in the body
10. Lifetime exposure to radiation in the workplace (i.e., being badged for radiation exposure), or exposure to radiation in the context of research protocol within the previous year that exceeds annual limits
11. More than one risk factor for coronary artery disease (e.g., smoking, hyperlipidemia, sedentary lifestyle)
12. Hypertension
13. Presence of clinically significant brain abnormalities. [For PET Scan Only]
14. Previous adverse reaction to stimulants that would preclude receiving methylphenidate
15. Presence or positive history of any cardiovascular disease, medical or neurological condition that would preclude methylphenidate administration or participation in this study
16. A history of bipolar disorder Type 1, or any history of syndromal psychosis
17. Lack of effective birth control

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 115 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2029-10-01 (Estimated); Study Completion 2030-10-01 (Estimated)

PRIMARY OUTCOMES:
Dopamine transmission | From the first (before methylphenidate) to the second PET scans (one hour after methylphenidate) on Day 1 of the study
  Delta BPND of [11C]raclopride in the Associative Striatum
Conversion to syndromal psychosis | From administration of the study drug to either conversion to a syndromal psychotic disorder or 24 months, whichever comes first.
  Development of a '6' on a P symptom of the SIPS

SECONDARY OUTCOMES:
Positive Symptoms | At time zero before administration of methylphenidate
  Total P symptom score on the SIPS
Negative Symptoms | At time zero before administration of methylphenidate
  Total N symptom score on the SIPS
Dopamine Transmission in the ventral striatum | From the first (before methylphenidate) to the second PET scans (one hour after methylphenidate) on Day 1 of the study
  Delta BPND ([11C]raclopride) in the Ventral striatum

OTHER OUTCOMES:
Baseline dopamine | At time zero before administration of methylphenidate
  Neuromelanin MRI in midbrain at baseline
Change in positive symptoms | From time zero before administration of methylphenidate to either conversion to a syndromal psychotic disorder or 24 months, whichever comes first.
  Change in total SIPS positive symptoms
Change in negative symptoms | From time zero before administration of methylphenidate to either conversion to a syndromal psychotic disorder or 24 months, whichever comes first.
  Change in total N symptoms on the SIPS

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared via the NIH data archive.
Time Frame: Data will be shared after the study has been completed, as per NIH guidelines.

REFERENCES:
- [Background] Girgis RR, Slifstein M, Brucato G, Kegeles LS, Colibazzi T, Lieberman JA, Abi-Dargham A. Imaging synaptic dopamine availability in individuals at clinical high-risk for psychosis: a [11C]-(+)-PHNO PET with methylphenidate challenge study. Mol Psychiatry. 2021 Jun;26(6):2504-2513. doi: 10.1038/s41380-020-00934-w. Epub 2020 Nov 5. PMID 33154566